CLINICAL TRIAL: NCT00571298
Title: A Phase I Trial of Extrapleural Pneumonectomy/Pleurectomy Decortication, Intrathoracic/Intraperitoneal Hyperthermic (IOHC) Cisplatin and Gemcitabine With Intravenous Amifostine and Sodium Thiosulfate Cytoprotection for Patients With Resectable Malignant Pleural Mesothelioma
Brief Title: Extrapleural Pneumonectomy /Pleurectomy Decortication, IHOC Cisplatin and Gemcitabine With Amifostine and Sodium Thiosulfate Cytoprotection for Resectable Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Raphael Bueno, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-091
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Extrapleural pneumonectomy; Pleurectomy Decortication; Mesothelioma; cisplatin; gemcitabine; amifostine; sodium thiosulfate
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Cisplatin; Gemcitabine; Amifostine; sodium thiosulfate; Cerebral Decortication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extrapleural pneumonectomy (EPP) (Experimental): This is dose escalation 3+3 study design. All the patients meet the eligibility criteria and then sign the informed consent. Then after they have completed their standard pre-operative evalutions were each brought to the operating room for this surgical resection. Regardless of the arm the subject is assigned to they all recieve surgical intervention (Extrapleural Pneumonectomy, Pleurectomy/Decortication, or Tumor Debulking), Amifostine, Cisplatin, Gemcitabine, and Sodium Thiosulfate
  Interventions: Procedure: Extrapleural pneumonectomy (EPP); Drug: Cisplatin; Drug: gemcitabine; Drug: amifostine; Drug: sodium thiosulfate
- Pleurectomy/Decortication (P/DC) (Experimental): This is dose escalation 3+3 study design. All the patients meet the eligibility criteria and then sign the informed consent. Then after they have completed their standard pre-operative evalutions were each brought to the operating room for this surgical resection. Regardless of the arm the subject is assigned to they all recieve surgical intervention (Extrapleural Pneumonectomy, Pleurectomy/Decortication, or Tumor Debulking), Amifostine, Cisplatin, Gemcitabine, and Sodium Thiosulfate
  Interventions: Drug: Cisplatin; Drug: gemcitabine; Drug: amifostine; Drug: sodium thiosulfate; Procedure: Pleurectomy/Decortication
- Tumor Debulking (TD) (Experimental): This is dose escalation 3+3 study design. All the patients meet the eligibility criteria and then sign the informed consent. Then after they have completed their standard pre-operative evalutions were each brought to the operating room for this surgical resection. Regardless of the arm the subject is assigned to they all recieve surgical intervention (Extrapleural Pneumonectomy, Pleurectomy/Decortication, or Tumor Debulking), Amifostine, Cisplatin, Gemcitabine, and Sodium Thiosulfate
  Interventions: Drug: Cisplatin; Drug: gemcitabine; Drug: amifostine; Drug: sodium thiosulfate

INTERVENTIONS:
Procedure: Extrapleural pneumonectomy (EPP) — Resection of the lung, the lining of the lung (pleura), the covering of the heart (pericardium), and the muscle that separates the chest and abdomen (diaphragm)
  Arms: Extrapleural pneumonectomy (EPP)
Drug: Cisplatin — Given after the tumor is removed as a bath (perfusion) for one-hour
  Other Names: Platinol
Drug: gemcitabine — Given after the tumor is removed as a bath (perfusion) for one-hour
  Other Names: Gemzar
Drug: amifostine — Given intravenously before perfusion chemotherapy and then 2 hours after the first dose
Drug: sodium thiosulfate — Given intravenously immediately at the end of perfusion chemotherapy
Procedure: Pleurectomy/Decortication — Resection of the lining of the lung (pleura), while the lung remains intact.
  Arms: Pleurectomy/Decortication (P/DC)

SUMMARY:
RATIONALE: After removal of visible cancer in the chest, chemotherapy drugs are used to kill or stop tumor cells from dividing, so that they stop growing or/and die. Cisplatin is currently used safely as in intra-operative treatment for malignant pleural mesothelioma. This study is aimed to determine if the addition of gemcitabine as a second intracavitary chemotherapy can be accomplished safely.

PURPOSE: This is a Phase I trial to study the efficacy of combination chemotherapy consisting of gemcitabine and cisplatin administered in the operating room and put into the chest and abdomen for one hour. We are also looking at the effects of heating the chemotherapy to a temperature of 42 degrees Celsius and the effect of cytoprotection agents: amifostine and sodium thiosulfate to counteract potential side effects of chemotherapy.

DETAILED DESCRIPTION:
* This is a dose escalation study of gemcitabine with a fixed dose of cisplatin
* Patients will undergo cytoreductive surgery, which entails the removal of the inner and outer lining of the lung (pleurectomy/decortication) with or without the lung itself (extrapleural pneumonectomy), including the lining overlying the pericardium and diaphragm. Resection of the pericardium and diaphragm are occasionally necessary to remove all visable tumor. This surgery is part of standard care for malignant pleural mesothelioma.
* After surgery, a one hour lavage with heated cisplatin and or gemcitabine will be administered to the hemithorax (and abdominal regions if the diaphragm is no longer present).
* Patients will remain hospitalized until they have recovered from surgery (usually 7-14 days).
* Patients will return to the hospital during the first month after their surgery to be evaluated by the medical staff.
* Dose escalation: 1) Three patients will be treated at the first dose level of gemcitabine. Labs will be monitored on a weekly basis, including a CBC, Chem-7, and LFT's. In the absence of developing dose-limiting toxicity (DLT) among the first 3 patients treated, dosages can be escalated. DLT will be defined as any grade 3 or higher renal toxicity, thrombocytopenia or other grade 3 toxicity not related to surgery 2) If none of these 3 patients have any toxicity, we will proceed to the next level of gemcitabine. 3) If DLT occurs in 1 of 3 patients at a given dose level, then 3 additional patients are added at that dose (for a total of 6 at this level)If no DLT occurs, we will proceed to the next level of gemcitabine. If DLT occurs in another patient, this dose is considered the maximum tolerated dose (MTD). 4) At any dose, 3 cases of DLT lead to discontinuation of recruitment at that dose and enrollment of 3 additional patients at a lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven diagnosis of stages I to III malignant mesothelioma of the pleura and negative mediastinal N2 lymph nodes (Malignancy is confined to the affected hemithorax)
* Adequate organ function including the following: adequate cardiac function, pulmonary function, renal and hepatic function and bone marrow reserve
* Adequate overall physical activity
* Surgical candidate for cytoreductive surgery

Exclusion Criteria:

* Extended disease outside the ipsilateral hemithorax as proven histologically, radiologically and/or intraoperatively
* Have received chemotherapy and or radiation therapy within the last 3 years at the time of study entry
* Serious concomitant systemic disorders
* Second active primary malignancy (to exclude non- melanoma skin cancer)
* Pregnancy at the time of the operation
* Psychiatric or addictive disorder which would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To establish the maximally tolerated dose (MTD) of intraoperative Intrathoracic/Intraperitoneal hyperthermic gemcitabine and cisplatin combination modulated by amifostine and sodium thiosulfate in patients with malignant pleural mesothelioma. | 2 years

SECONDARY OUTCOMES:
To determine and quantitate the safety of this combination in these patients by defining the dose limiting toxicity. | 2 years
To study the pharmacokinetics of gemcitabine and cisplatin combination administered in this way. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Brigham and Women's Hospital, Mesothelioma and International Mesothelioma Program — http://www.brighamandwomens.org/mesothelioma